CLINICAL TRIAL: NCT00882180
Title: A Multi-Center, Open Label, Phase 1 Dose-Escalation Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous ALN-VSP02 in Patients With Advanced Solid Tumors With Liver Involvement
Brief Title: Dose Escalation Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous ALN-VSP02 In Patients With Advanced Solid Tumors With Liver Involvement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-VSP02-001
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Solid Tumors
Keywords: Liver; Solid Tumors; Advanced Solid Tumors with Liver Involvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ALN-VSP02 — IV infusion administered every two weeks

SUMMARY:
The purpose of the study is to determine the safety, tolerability, pharmacokinetics, and pharmacodynamics of intravenous ALN-VSP02, an RNAi therapeutic, in patients with advanced solid tumors with liver involvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced solid tumors that have recurred or progressed following standard therapy, or that have not responded to standard therapy, or for which there is no standard therapy, or who are not candidates for standard therapy
* Patient has measurable tumor in the liver
* At least 28 days have elapsed since the patient's prior systemic therapy, radiotherapy, or any major surgery
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1
* Patient has adequate hematologic, liver, and renal function
* Patient is seronegative for hepatitis B virus (HBV) and hepatitis C virus (HCV)
* Patient has a life expectancy > 12 weeks

Exclusion Criteria:

* Patient is receiving full-dose (therapeutic) anticoagulation therapy and/or aspirin > 325 mg/day or other platelet inhibitory agents
* Patient has clinically significant cardiovascular disease or uncontrolled serious cardiac arrythmia
* Patient has known active brain or leptomeningeal metastases
* Patient has clinically significant cerebrovascular disease
* Patient has a seizure disorder not controlled on medication
* Patient has a known or suspected viral, parasitic or fungal infection
* Patient previously experienced a severe reaction to a liposomal product
* Patient has a known hypersensitivity to lipid products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of intravenous ALN-VSP02 | up to 16 weeks (4 cycles)

SECONDARY OUTCOMES:
Plasma and urine PK of ALN-VSP02 | 8 weeks (two cycles)
Assess preliminary evidence of antitumor/antiangiogenic activity | Up to 16 weeks (4 cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Vaishnaw, MD PhD, Study Director — Alnylam Pharmaceuticals
Locations (10):
- United States (7):
  - TGen Clinical Research Service at Scottsdale Healthcare, Scottsdale, Arizona
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Spain (3):
  - Hospital Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Vall d'Hebron, Barcelona, Catalonia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia